CLINICAL TRIAL: NCT01674660
Title: Factors Associated With Interdialytic Blood Pressure Variability in Maintenance Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Ma Weihua, Principal Investigater, Beijing Chao Yang Hospital
Other Study IDs: BeijingCYH; 19860805 (Registry Identifier: Ma Weihua)
Record Dates: First submitted 2012-08-21; First posted 2012-08-29 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Kidney Failure, Chronic
Keywords: hemodialysis; blood pressure variability; volume status
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine.

GROUPS / COHORTS (3):
- volume status: volume status:group1 over volume status,group2 normal volume status,group3 low volume status
- night blood pressure: night blood pressure：group1 nondipper,group2 dipper,group3 extreme dipper,group4 riser
- interdialysis weight gain: interdialysis weight gain:group1 >5% dry weight,group2 <5% dry weight

SUMMARY:
The purpose of this study is to explore the factors associated with interdialytic blood pressure variability in maintenance hemodialysis patients, especially the association between volume status and blood pressure variability.

DETAILED DESCRIPTION:
Hemodialysis patients experience higher rates of cardiovascular morbidity and mortality than the general population and many populations with other chronic diseases. This exceptional risk is explained in part by known risk factors such as diabetes, hypertension, and other uremia-related factors, including vascular calcification and stiffness, autonomic dysfunction, and a high burden of circulating inflammatory mediators. However, additional unidentified risk factors also likely contribute to the disproportionately high prevalence of cardiovascular morbidity in hemodialysis patients. Blood pressure variability may represent one plausible cardiovascular risk factor. Data from nonuremic human populations show an association between greater blood pressure variability and cardiovascular events,nonfatal cardiovascular events,stroke,and increased left ventricular mass. There has been comparatively little work examining the causes and effects of blood pressure variability in hemodialysis populations. So the purpose of this study is to explore the factors associated with interdialytic blood pressure variability in maintenance hemodialysis patients, especially the association between volume status and blood pressure variability.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* receipt of thrice-weekly in-center hemodialysis
* no anticipation of imminent(<6 months)living related kidney transplant
* not transfer of care to a nonparticipating facility
* no dialytic modality change
* free of vascular, infectious, or bleeding complication within 1 month Exclusion Criteria:
* who missed >2 hemodialysis treatments over 1 month
* abused drugs
* severe anemia，malnutrition，chronic atrial fibrillation
* body mass index of 40 >kg/m2

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients of Beijing Chaoyang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
interdialytic blood pressure | 44 hours
  Ambulatory BP monitoring was performed after the midweek hemodialysis session for 44 hours. Ambulatory BPs were recorded every 20 minutes during the day (6 AM to 10 PM) and every 30 minutes during the night (10 PM to 6 AM) in the nonaccess arm, We use the coefficient of variation or standard deviation in interdialytic blood pressure as a indicator of systolic blood pressure variability.

CONTACTS AND LOCATIONS:
Overall Officials: Ma WH weihua, Master, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Nephrology, dialysis center,Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China